CLINICAL TRIAL: NCT06172166
Title: Transdisciplinary Care for Young Adults With Type 1 Diabetes Transitioning to Adult Healthcare
Brief Title: Transdisciplinary Care for Young Adults With Type 1 Diabetes
Acronym: TCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Albert Einstein College of Medicine (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Jessica Pierce, Senior Research Scientist, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JDRF_TCT
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transdisciplinary Care for Transition (Experimental)
  Interventions: Behavioral: Transdisciplinary Care for Transition
- Standard Clinical Care (No Intervention)

INTERVENTIONS:
Behavioral: Transdisciplinary Care for Transition — Young adults with T1D will participate in three visits during which they will see a diabetes nurse educator, psychologist, and transition navigator/social worker who will co-deliver care. TCT Visits 1 and 2 will be before the first adult diabetes healthcare visit, during trial months 1 and 2 respectively. These visits will focus on improving transition readiness, establishing care with an adult T1D specialist, and navigating psychosocial barriers to successful transition. TCT Visit 3 will occur after the first adult T1D healthcare visit, within one month of the first adult T1D care visit or during trial month 7 if the visit has not yet occurred. TCT Visit 3 will focus on overcoming barriers to satisfactory adult T1D healthcare.
  Arms: Transdisciplinary Care for Transition

SUMMARY:
The incidence of type 1 diabetes (T1D) is increasing globally with the most substantial increases occurring in the youngest age groups. A growing number of youths with T1D must therefore transition their healthcare from pediatric to adult T1D care settings as they approach young adulthood. This healthcare transition introduces many challenges because it coincides with a developmental period that is fraught with social, financial, residential, school/work and other changes/demands. Thus, it is not surprising that young adults (YA) with T1D are at risk for suboptimal glycemic levels, the development of diabetes-related complications, and psychosocial issues such as depression, anxiety, and disordered eating. Yet, few evidence-based interventions to assist YA with T1D with this complex healthcare transition exist.

In this study, we are testing the feasibility, acceptability, and initial efficacy of a novel transdisciplinary model of care (Transdisciplinary Care for Transition; TCT) in which a diabetes nurse educator, psychologist, and transition navigator (case manager) co-deliver transitional care. TCT addresses the psychological and systems barriers to transition and aims to improve outcomes via better assessment of YA needs and resources, better cross-discipline and YA-provider communication, and better collaboration with YA to resolve problems that cross pediatric and adult healthcare settings.

We will recruit 80 YA with T1D during their final visit in pediatric T1D specialty care to participate in a pilot randomized controlled trial during which we will randomize YA to a standard care control group (SCC) or to receive three TCT visits during the 6 months post discharge from pediatric T1D care. In SCC, participants will transition to adult T1D care as usual per their clinic's standard transition procedures.

All study procedures can be completed remotely. This includes enrollment, study evaluations, and TCT visits for those randomized to TCT. Thus, we are recruiting individuals from across the United States.

Aim 1: Examine the feasibility, acceptability, and fidelity of TCT in YA with T1D.

Aim 2: Examine the preliminary efficacy of TCT versus SCC on YA HbA1c, transition readiness and success, and continuity of care and explore for an effect on diabetes distress and acute care utilization.

DETAILED DESCRIPTION:
All study procedures can be completed remotely. This includes enrollment, study evaluations, and TCT visits for those randomized to TCT. Thus, we are recruiting individuals from across the United States.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes for at least 6 months
* Approaching their last visit with their pediatric type 1 diabetes healthcare provider. They will have their final visit with their pediatric T1D provider within about a month of enrollment in the study.
* English fluency

Exclusion Criteria:

* Another systemic chronic medical illness except celiac disease, autoimmune thyroiditis, microalbuminuria, hypertension, or well-managed asthma
* Developmental disability limiting independent living

We are recruiting eligible individuals through Nemours and remotely.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic level | Baseline, 6-months, 12-months
  HbA1c via mailed dried blood spot (DBS) kits
Transition readiness | Baseline, 6-months, 12-months
  Readiness Assessment of Emerging Adults with Type 1 Diabetes Diagnosed in Youth (READDY): self-report of confidence of T1D health knowledge and skills needed for transition.
Transition outcomes | 6-months, 12-months
  Healthcare Transition Outcomes Inventory (HCTOI): self-report of perceived level of success on multiple dimensions of healthcare transition outcomes
Time to First Adult Care Visit | 6-months, 12-months
  Self-report and medical record review of the time between the last pediatric T1D care visit and the first adult T1D care visit
Continuity of care | 6-months, 12-months
  Self-report and medical record review of the number of visits in adult T1D care since last study visit

SECONDARY OUTCOMES:
Diabetes distress | Baseline, 6-months, 12-months
  Diabetes Distress Scale for Adults with T1D (T1-DDS): self-report of emotional distress associated with the ongoing worries, burdens, and concerns of living with T1D
Acute care utilization | 6-months, 12-months
  Self-report and medical record review of the number of T1D-related emergency department visits, urgent care visits, and hospital admissions (and reason why) since last study visit
Level 3 (Severe) Hypoglycemia | 6-months, 12-months
  Self-report and medical record review of the number of severe hypoglycemic events characterized by altered mental status and/or physical status requiring assistance since last study visit
Diabetic Ketoacidosis | 6-months, 12-months
  Self-report and medical record review of the number of episodes of DKA since last study visit.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nemours Children's Health, Delaware, Wilmington, Delaware
  - Nemours Children's Health, Florida, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No